CLINICAL TRIAL: NCT03922256
Title: Prospective, Observational Clinical Investigation of the Exos® Reformable Brace for Conservatively Managed Distal Radius Fractures: An Evaluation of Time to Union, Satisfaction, and Convenience
Brief Title: Prospective, Observational Clinical Investigation of the Exos Reformable Brace
Acronym: EXOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: Encore DJO Global (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FORE EXOS Brace 2018
Record Dates: First submitted 2019-02-13; First posted 2019-04-19 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: This single-cohort, consecutive series clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brace Arm (Experimental): All subjects in this study received the reformable brace
  Interventions: Other: molded brace

INTERVENTIONS:
Other: molded brace — The moldable brace utilized in the current study will be pre-fabricated and of the short-arm brace variety , which is primarily indicated for non-displaced fractures of the distal radius or distal ulna. The braces are available in multiple sizes for both right and left hands.

SUMMARY:
This is a prospective observational single cohort trial quantifying time to radiographic union (primary endpoint) and convenience, satisfaction, pain and resource requirements (secondary) for patients with non-operatively treated distal radius fractures managed with a thermoformable Exos short-arm brace.

DETAILED DESCRIPTION:
The trial will be a prospective trial of a convenience sample of skeletally mature patients with radiographically-confirmed distal radius fractures that can be managed without ORIF. The study population will be defined as all adult patients (>18 years) with stable, non-displaced distal radius fractures. All patients will be independent in activities of daily living. Patients will be screened as candidates for enrollment into the study and if the patient satisfies the inclusion/exclusion criteria, a clinical research coordinator or the study PI/coPI will explain all essential elements of the clinical trial. If the patient agrees to participate, the study coordinator or PI/coPI will obtain informed consent. The patient will still be followed clinically per the PI/coPI's standard of care.

ELIGIBILITY:
Inclusion

* Age > 18 years;
* Unilateral fracture of distal radius without misalignment (dorsal angulation <10°, axial radial shortening <5mm), <2mm intraarticular stepoff;
* Independent in activities of daily living;
* Capable and willing of signing informed consent.

Exclusion

* Children under the age of 18;
* Fracture of the contralateral arm;
* Other fractures of the ipsilateral arm;
* Open fractures;
* Fractures that require reduction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
bony union | 2-12 weeks
  radiographic time to union

SECONDARY OUTCOMES:
Patient Reported Outcomes | 2-12 weeks
  Visual Analog Scale from 1(no pain) to 100(extreme pain)
Patient Reported Disability Scale- Quick-DASH | 2-12 weeks
  11 questions rating ability of activites - ranging from no difficulty to unable to do
Patient rated Wrist Evaluation | 2-12 weeks
  Rates pain and function on 1(no pain) to 10 (worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Nydick, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States